CLINICAL TRIAL: NCT04950673
Title: Open-label, Post-marketing, Prospective, Two-Armed Comparison Study to Assess Impact of SARS-CoV-2 or COVID-19 on Cognitive Function in Patients
Brief Title: Open-label, Post-marketing, Prospective Study to Assess Impact of COVID-19 on Cognitive Function in Patients
Acronym: COVID19
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cognivue, Inc. (Industry)
Collaborators: Kaweah Delta District Hospital (Unknown); Riiid Research LLC (Unknown); UH, Cleveland Medical Center (Unknown); US Medical Care INC (Unknown)
Responsible Party: Sponsor
Other Study IDs: COG-COVID19
Record Dates: First submitted 2021-06-30; First posted 2021-07-06 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Cognitive Decline; Cognitive Dysfunction; Brain Health; Post CoV-2 Syndrome; COVID Long-Haul
Keywords: SARS-CoV2; COVID19; Cognition; Cognivue; Institutional Review Board or IRB; Montreal Cognitive Assessment or MoCA; Mini-Mental Status Exam or MMSE; Patient Health Questionnaire or PHQ-9; Food Drug Administration or FDA; World Health Organization or WHO; Informed Consent Form or ICF; Case Report Form or CRF; Good Clinical Practice or GCP; Post CoV-2 Syndrome; COVID Long-Haul
MeSH Terms: conditions — Cognitive Dysfunction; Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Subjects who had COVID-19 infection and recovered at 3 months: 500 subjects who have had a history of COVID19 infection and recovered 3 months prior to the enrollment
  Interventions: Device: Cognivue
- Subjects who never had COVID-19 infection: 500 subjects who never had a history of COVID19 infection prior to the enrollment
  Interventions: Device: Cognivue

INTERVENTIONS:
Device: Cognivue — Computerized Cognitive Assessment Device

SUMMARY:
The objective of this study is to compare the impact of the coronavirus disease (SARS-CoV-2, or COVID-19) on cognitive function in the population of patients who have been diagnosed, treated and recovered from the COVID-19 infection versus patients who have not been infected. Primary endpoint is to evaluate the percentage of cognitive decline observed in both study arms (subjects with or without COVID-19 history) using assessments of Cognivue Clarity, MMSE and MoCA. Secondary endpoint is to see the correlation of Depression and anxiety scales (i.e., Patient Health Questionnaire-9 (PHQ-9) and/or Geriatric Depression Scale (GDS)) and Cognivue scores while comparing the trend of difference between both study arms.

DETAILED DESCRIPTION:
Cognivue is an FDA-cleared cognitive assessment device based on modern cognitive neuroscience, that allows physicians, allied healthcare providers, and patients to access a new approach to brain health, moving beyond the old questions and answers approach of traditional cognitive tests.

Cognivue's development and testing is based on 20 years of psychophysical and neurophysiological research that has focused on the early detection of patients' cognitive decline. Its FDA clearance study demonstrated significant correlation to the SLUMS and other neuropsychological tests, superior test re-test reliability compared to SLUMS, and validated its psychometric properties.

Historically, physicians have used the Mini-Mental Status Exam (MMSE) and Montreal Cognitive Assessment (MoCA) to assess cognitive functioning. These tools are often limited by issues of bias, inconsistent retest reliability, staffing and cost. The automated Cognivue technology utilizes adaptive psychophysics and assesses the patient's motor skills and visual acuity, eliminating the bias found in common cognitive testing mechanisms such as MMSE, MoCA, and Mini-Cog.

Using Cognivue Clarity, we have an opportunity to better understand a person in total when we insist that cognitive function testing is part of the recovery plan for individuals who experience the whiplash of COVID-19, either directly or indirectly.

This is a multi-site, open-label study. Approximately 1000 subjects will be enrolled. Up to 500 subjects with COVID-19 history and 500 subjects without a COVID-19 diagnosis will be enrolled in this study.

During the first visit, all subjects will be provided with an informed consent form (ICF) to review and sign prior to starting any study-specific procedures. Subjects will be asked about their COVID-19 diagnosis history, prior to study enrollment. After informed consent is obtained from subjects, study staff will review contact, demographic and medical history information. Following this review, cognitive testing using Cognivue Clarity, MMSE and MOCA will occur. In addition, subjects will take the Patient Health Questionnaire-9 (PHQ-9) and/or Geriatric Depression Scale (GDS) during this visit .

Subjects will be followed for 24 months in the study, coming to the study site to review COVID-19 infection (re-infection or newly diagnosed) as well as perform cognitive testing with Cognivue Clarity, MMSE and MOCA. Subjects will also take the PHQ-9 and/or GDS during these visits. In addition, during the 12- and 24-month visits, study staff will review previously reported medical history information with subjects to determine any new information.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Male or Female
* Previous diagnosis of COVID-19, but recovered >3 months (Arm 1)
* Never infected or diagnosed with COVID-19 (Arm 2)
* Fluent in English
* Able to operate simple computerized device
* Willing to sign a written informed consent and ability to comply with study requirements
* Ability to provide demographic and medical history information

Exclusion Criteria:

* Individuals under 18 years old
* Currently under COVID-19 treatment or quarantine
* Previously known diagnosis of dementia and Alzheimer's
* Inability to provide written informed consent for self or complete cognitive testing (either using Cognivue Clarity or paper/pencil testing)
* Known severe terminal illness

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — males and females
Study Population: 1000 total subjects; 500 with COVID-19 history and 500 without COVID-19 diagnosis.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive decline | 24 months
  The percentage of cognitive decline observed in both study arms (subjects with or without COVID-19 history) using assessments of Cognivue Clarity, Mini Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA).

SECONDARY OUTCOMES:
Comparison between Cognivue and other paper-pencil cognitive assessment batteries | 24 months
  Depression and anxiety scales, i.e., Patient Health Questionnaire-9 (PHQ-9) or Geriatric Depression Scale (GDS).

CONTACTS AND LOCATIONS:
Overall Officials: Diego Cahn-Hidalgo, MD, Principal Investigator — Cognivue, Inc.
Locations (4):
- United States (4):
  - RiiiD Research, LLC, Irvine, California
  - Kaweah Health (Kaweah Delta District Hospital), Visalia, California
  - US Medical Care Inc, Boca Raton, Florida
  - UH Cleveland Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
No plan to share participants' data with other researchers due to the HIPAA compliant issue